CLINICAL TRIAL: NCT04679207
Title: A Pilot Study of Ultrasound-guided Vacuum-assisted Excision of Breast Cancers (the PICASSO Study)
Brief Title: A Pilot Study of Ultrasound-guided Vacuum-assisted Excision of Breast Cancers
Acronym: PICASSO
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00157
Record Dates: First submitted 2020-11-25; First posted 2020-12-22 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participant will be given the option to consent to donating any surplus tumour tissue for use in other ethically approved studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Vacuum-assisted excision — Vacuum-assisted biopsy (VAB) is a minimally invasive technique performed under local anaesthetic as an outpatient procedure by radiologists using x-ray or ultrasound guidance. It was developed in the USA in the mid 1990s and has become well established as a diagnostic test for suspected breast disease. It uses the combination of a large gauge biopsy needle and suction to allow larger pieces of tissue to be removed than can be obtained with a standard needle biopsy device. The technique is used widely for diagnostic purposes and, in some centres, for the therapeutic removal of benign breast lumps such as fibroadenomas and papillomas.

SUMMARY:
This study is looking into whether the procedure called Vacuum Assisted Excision (VAE) is a safe method for the removal of small and medium sized invasive breast cancers in patients who are unfit or have refused to have surgery to remove cancer.

Recruitment Target: 20

ELIGIBILITY:
Inclusion Criteria:

* The patient is aged 18 years or older.
* Diagnosis on core needle biopsy of invasive cancer of the breast
* Unifocal invasive tumour on imaging (hormone receptor positive or negative)
* T1 or T2 primary or locally recurrent tumour measuring ≤25mm on imaging, excluding any adjacent ductal carcinoma in situ (largest of the measurements on mammography (including digital breast tomosynthesis if performed) and ultrasound)
* The tumour is clearly visible on ultrasound
* Vacuum-assisted excision of the entire ultrasonically visible tumour is deemed to be technically feasible
* The patient is considered to be at high risk of complications or death from a general anaesthetic and therefore surgery under general anaesthesia is not considered appropriate. This must be confirmed by agreement by two named consultant breast surgeons, a multidisciplinary team meeting (including at least one consultant breast surgeon) or by formal anaesthetic assessment. Unsuitability for surgery under local anaesthetic must be confirmed by a consultant breast surgeon.
* or - The patient refuses to undergo surgery. This must be confirmed by a consultant surgeon and breast care nurse following full discussion of the treatment options.
* or - The patient is considered unlikely to benefit from surgical removal of the cancer by virtue of known metastatic disease or other life-shortening condition. This must be confirmed by discussion in a multidisciplinary team meeting which includes an oncologist.
* The patient has given written informed consent for the study Women who are already on primary endocrine therapy for a breast cancer and meet the inclusion criteria will also be eligible.

Exclusion Criteria:

* The patient is on anticoagulants or has a known clotting disorder
* Pregnancy or lactation
* Allergy to local anaesthetic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who require a safe method for the removal of small and medium sized invasive breast cancers in patients who are unfit or have refused to have surgery to remove cancer.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Greatest dimension of the Cancer | 1 year
  The proportion of participants in whom the greatest dimension of the cancer on imaging at 1 year post-vacuum assisted excision (VAE) is ≤50% of its pre-VAE size.

SECONDARY OUTCOMES:
Recruitment Uptake | 12 months
  Proportion of eligible women offered the study who consent to participate.
Procedure Times | 12 months
  Time taken for each VAE procedure.
Procedure pain and acceptability | 12 months
  11-point numerical rating pain score - with 0 being no pain and 10 being worst pain imaginable
Complication rate of VAE | 12 months
  Proportion of women who have significant bleeding after the procedure (defined as bleeding requiring > 20 minutes manual compression to control and/or a haematoma requiring aspiration or surgical evacuation) or infection at the VAE site (defined as requiring antibiotic treatment and/or an abscess requiring aspiration or surgery).
Proportion of Cancer removed | 12 months
  Proportion of women in whom the cancer appears to be completely removed as judged on ultrasound at the end of the VAE procedure
Residual Cancer after VAE | 2 years post VAE
  Proportion of participants in whom the greatest dimension of the cancer on imaging at 2 years post-VAE is less ≤ 50% of its pre-VAE size.
Requirement of salvage surgery | 2 years post VAE
  Proportion of participants who undergo surgery to the ipsilateral breast within 2 years of the VAE procedure because of continued growth of the tumour.
Histopathology of cavity walls | Imaging at 1 year and 2 years.
  Proportion of participants with positive and negative cavity wall biopsies respectively who have tumour visible on imaging at 1 and 2 years.
proportion willing to undergo the procedure again if necessary. | 12 months
  proportion willing to undergo the procedure again if necessary based on yes or no question

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom